CLINICAL TRIAL: NCT03395483
Title: Investigating the Peripheral Perfusion Index; Correlations Between Peripheral and Mesenteric Perfusion in Elective Surgical Patients
Brief Title: Peripheral and Mesenteric Perfusion in Elective Surgical Patients
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Højlund, MD, Senior Hospital Physician, Hvidovre University Hospital
Other Study IDs: H-17004663
Record Dates: First submitted 2017-12-16; First posted 2018-01-10 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Perfusion; Bowel Ischemia; Colorectal Surgery; Haemodynamic Instability
Keywords: peripheral perfusion; Haemodynamic Instability; mesenteric bloodflow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective, adult colorectal surgical patients: All patients will be monitored by the non-invasive Masimo Radical7 pulseoximeter (Masimo, Irvine, CA, USA) measuring PPI and the MoorVMS-LDF (Moor Instruments Ldt., Axminster, UK) measuring mesenteric tissue blood flow using doppler flowmetry. Patients will be subjected to a haemodynamic challenge using anti-trendelenburg position.
  Interventions: Other: Haemodynamic monitoring

INTERVENTIONS:
Other: Haemodynamic monitoring — see Group description

SUMMARY:
An important goal of haemodynamic monitoring and resuscitation is early detection of insufficient tissue perfusion and oxygenation. The mesenteric haemodynamic response to circulatory shock is complex, and diagnosis of bowel ischaemia poses significant difficulty. Assuming blood flow is diverted from the peripheral tissue and the gastrointestinal tract to vital organs, during circulatory shock, an objective, simple and non-invasive method of detecting peripheral tissue perfusion impairment might detect this at an early stage.

The peripheral perfusion index (PPI) reflects changes in peripheral perfusion and laser doppler flowmetry allows measurement of bowel tissue perfusion.

The aim of this study is to explore the association between changes in peripheral and intestinal perfusion in patients undergoing elective colorectal surgery exposed to intraoperative haemodynamic challenges.

DETAILED DESCRIPTION:
An important goal of haemodynamic monitoring and resuscitation is early detection of insufficient tissue perfusion and oxygenation, but in clinical practice, monitoring and resuscitation is routinely based on measuring of blood pressure and heart rate, which might be inadequate endpoints for optimal resuscitation. Haemodynamic management targeting cardiac output and stroke volume (SV), and to some extent, flow and tissue perfusion is feasible when applying minimally-invasive or non-invasive methods, but has been limited to a narrow number of critically ill patients and to the intraoperative setting. Another approach to resuscitation is aimed at flow and perfusion of vital organs. Ideally, measurements would be done directly on these organs, but no feasible methods exist. Assuming blood flow is diverted from the peripheral tissue and the gastrointestinal tract to vital organs, during circulatory shock, an objective, simple and non-invasive method of detecting peripheral tissue perfusion impairment might detect this at an early stage. The peripheral perfusion index (PPI) is derived from the photoelectric plethysmographic pulse oximetry signal, which all patients are monitored by perioperatively to assess arterial oxygen saturation. The PPI is a numerical non-invasive measure representing the ratio between the pulsatile (arterial) and non-pulsatile component of the light reaching the pulse oximeter, and PPI decreases in states of hypoperfusion. PPI reflects changes in peripheral perfusion and blood volume and decreased peripheral perfusion determined by PPI predicts surgical complications and morbidity in acute surgical and septic shock patients.

The mesenteric haemodynamic response to circulatory shock is complex, and diagnosis of bowel ischaemia poses significant difficulty for the clinicians due to its non specific presentations and lack of a simple diagnostic test. In patients undergoing colorectal surgery for malignancy, laser doppler flowmetry allows measurement of bowel tissue perfusion.

The aim of this study is to explore the association between changes in peripheral and intestinal perfusion in patients undergoing elective colorectal surgery exposed to intraoperative haemodynamic challenges.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Elective colorectal surgery, low anterior resection of the colon, sigmoid colectomy or right hemicolectomy
* Written informed consent

Exclusion Criteria:

* No consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: x
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Peripheral perfusion index and mesenteric perfusion changes from baseline after haemodynamic challenges | Perioperatively
  Association between PPI and mesenteric perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Agerskov, MD, Research Fellow, Study Chair — Department af Anaesthesia, Hvidovre Hospital, University of Copenhagen; Jakob Højlund, Chief Physician, Principal Investigator — Department of Anaesthesia, Hvidovre Hospital, University of Copenhagen; Nicolai Bang Foss, Clinical Professor, DMSc., Study Director — Department of Anaesthesia, Hvidovre Hospital, University of Copenhagen; Henrik Sørensen, MD, DMSc., Study Chair — Department of Anaesthesiology, Abdominal Centre, Rigshospitalet, University of Copenhagen; Niels Secher, Professor, DMSc., Study Chair — Department of Anaesthesiology, Abdominal Centre, Rigshospitalet, University of Copenhagen
Locations (1):
- Anæstesiologisk afdeling, Hvidovre hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No